CLINICAL TRIAL: NCT01381341
Title: A Phase 1 Pharmacokinetic Study To Compare the Relative Bioavailability of Two Clinical Formulations of Linifanib in Subjects With Solid Tumors
Brief Title: To Compare Relative Bioavailability of Two Clinical Formulations of Linifanib.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M11-817
Record Dates: First submitted 2011-06-14; First posted 2011-06-27 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- linifanib (Experimental)
  Interventions: Drug: linifanib

INTERVENTIONS:
Drug: linifanib — QD on Day 1 of Periods 1 and 2
  Other Names: ABT-869

SUMMARY:
A pharmacokinetic study to compare 2 clinical formulations of linifanib.

DETAILED DESCRIPTION:
This study is designed to evaluate the bioavailability of linifanib from 2 formulations. Subjects may enroll in a separate extension study to continue receiving linifanib after completion of this study.

ELIGIBILITY:
Inclusion Criteria

1. Age is greater than or equal to 18 years.
2. Subject must have a histologically or cytologically confirmed non-hematologic malignancy other than Hepatocellular Carcinoma (HCC).
3. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
4. Subject must have adequate bone marrow, renal and hepatic function as follows:

   * Bone Marrow: Absolute neutrophil count (ANC) >= 1,500/mm^3 (1.5 X 10^9/L); Platelets >= 75,000/mm^3 (75 X 10^9/L); Hemoglobin >= 9.0 g/dL (1.4 mmol/L)
   * Renal function: serum creatinine <= 2.0 mg/dL (0.81 mmol/L);
   * Hepatic function: AST and ALT <= 1.5 X ULN unless liver metastases are present, then AST and ALT <= 5.0 X ULN; bilirubin <= 1.5 mg/dL (0.026 mmol/L)
5. Subject must have Partial Thromboplastin Time (PTT) </= 1.5 x Upper Limit of Normal ( ULN) and International Normalized Ratio (INR) </= 1.5.

Exclusion Criteria

1. Subject has received anti-cancer therapy including investigational agents, cytotoxic chemotherapy, radiation therapy or biologic therapy within 21 days or within a period defined by 5 half lives, whichever is shorter, prior to study drug administration. In addition subject has not recovered to less than or equal to Grade 1 clinically significant adverse effects/toxicities of the previous therapy.
2. Subject has undergone major surgery within 21 days of Period 1, Study Day 1.
3. Subject has untreated brain or meningeal metastases. Subjects with treated brain metastases that are radiographically or clinically stable (for at least 4 weeks after therapy) and who have no evidence of cavitation or hemorrhage in the brain lesion, are eligible provided that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to Study Day 1, Period 1).
4. Current enrollment in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetic profile of linifanib in subjects with advanced or metastatic solid tumors. | At various time points from Day 1 through Day 5 of Periods 1 and 2
  Blood samples for the pharmacokinetics (PK) of linifanib will be collected at designated time points and assayed.

SECONDARY OUTCOMES:
Safety: Adverse Events - The number of participants with adverse events will be reported as a measure of Safety. | Throughout the study
  The investigators will monitor each subject for clinical and lab evidence of adverse events on a routine basis through out the study.
Safety: Physical Examination and Vital Signs - Physical examination will be performed and vital signs will be assessed for participants as a measure of safety. | Physical exam at Screening, Day 1 of Periods 1 and 2 and Day 5, Period 2/Final Visit and 30 day safety follow-up; Vital Signs (blood pressure, heart rate, body temperature) will be done at all visits.
  Complete physical exam, including body weight, will be done at Screening. A symptom-directed physical exam, including bodyweight, will be done at Day 1, Periods 1 and 2, Day 5, Period 2/Final Visit and 30 day safety follow-up.
Safety: Clinical Lab Tests will be performed for each participant as a safety measure. | Screening, Day 1, Periods 1 and 2, Day 5, Period2/Final Visit and 30 day safety follow-up.
  Chemistry, hematology, urinalysis lab tests

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. McKee, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 51403, Tacoma, Washington, United States